CLINICAL TRIAL: NCT04545528
Title: The Impact of Nutritional Service in the Stone Clinic on the Patient Urine
Brief Title: The Impact of Nutritional Service in the Stone Clinic on the Patient Urine Collection Results
Acronym: NUT1
Status: Withdrawn | Type: Observational
Why Stopped: Logistical problems in clinic
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ilan Beniamin Klein, Principal investigator, Carmel Medical Center
Other Study IDs: CMC-20-0013-CTIL
Record Dates: First submitted 2020-08-25; First posted 2020-09-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Kidney Stone; Kidney Calculi
Keywords: kidney stone; kidney Caliculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: 100 Patients that were referred to our stone clinic for follow up with risk factors for stone recurrence like metabolic syndrome and diabetes, uric acid stones etc. In addition to seeing our urologist and nephrologist these patients will also be referred to a nutritionist in order to balance risk factors and will be followed for one year with our usual blood tests and imaging
  Interventions: Behavioral: Dietary recommendations
- Control group: 100 Patients that were referred to our stone clinic for follow up without risk factors for stone recurrence will see our urologist and nephrologist and will be followed for one year with our usual blood tests and imaging

INTERVENTIONS:
Behavioral: Dietary recommendations — The test group will be seen by a nutritionist and will receive specific dietary recommendations according to their specific comorbidities and drugs
  Groups: Test group

SUMMARY:
Kidney stone disease has become a common phenomenon in the US and Europe with a growing incidence of about 10%. Life style and dietary changes have a cardinal part in kidney stone prevention. Therefore it was only natural to determine the impact of the addition of a nutritionist to a stone clinic run by a urologist and a nephrologist.

DETAILED DESCRIPTION:
Kidney stone disease has become a common phenomenon in the US and Europe with a growing incidence of about 10%. A history of kidney stone disease has also been connected to cardiovascular and renal insufficiency events to a point that kidney stones is looked at today as a systemic predictor of hypertension, cardiovascular disease and more.

Seeing the importance of these risk factors we initiated a stone clinic for our kidney stone patients several years ago run jointly by a urologist and a nephrologist. Seeing that life style and dietary changes have a cardinal part in kidney stone prevention, it was only natural to determine the impact of the addition of a nutritionist to a stone clinic run by a urologist and a nephrologist on our patient parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18 yo and older
* 2 kidneys
* Kidney or ureteric stone treated surgically or conservatively

Exclusion Criteria:

* Single kidney
* Aberrant kidney anatomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients18 yo and older referred to out kidney stone clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
24h Urine collection results | Through study completion, an average of 1 year
  to follow changes in the 24 hour urine collection results that are routinely taken as part as follow up: volume in millilitres; calcium, oxalate, magnesium, phosphorus sodium and potassium in mg/day;

SECONDARY OUTCOMES:
Weight | Through study completion, an average of 1 year
  weight in kilograms
Height | Through study completion, an average of 1 year
  Height in meters
BMI | Through study completion, an average of 1 year
  Calculated BMI using the above weight and height
Creatinin in mg/dl | Through study completion, an average of 1 year
  Lab results
Calcium in mg/dl | Through study completion, an average of 1 year
  Lab results
sodium in mg/dl | Through study completion, an average of 1 year
  Lab results
potassium in mg/dl | Through study completion, an average of 1 year
  Lab results

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Lady Davis Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided